CLINICAL TRIAL: NCT07222722
Title: Near Infrared Spectroscopy (NIRS) Monitoring as an Early Predictor of Acute Kidney Injury (AKI) in a Vulnerable Neonatal Intensive Care Unit (NICU) Population
Brief Title: NIRS Monitoring in the NICU and AKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-00172
Record Dates: First submitted 2025-10-29; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Acute Kidney Injury (AKI); Postnatal AKI
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- NICU patients born less than 30 weeks gestational age (Experimental): All patients included in the study will be assigned to receive NIRS monitoring.
  Interventions: Device: NIRS Monitoring

INTERVENTIONS:
Device: NIRS Monitoring — The renal NIRS device is a non-invasive tool that uses near-infrared light to measure oxygen saturation various tissues. Renal NIRS sensors will be placed by 24 hours of the participants' admission.

SUMMARY:
The primary objective of this study is to describe the pattern of renal tissue oxygen saturation (SrSO2) using near-infrared spectroscopy (NIRS) in premature infants <30 weeks gestational age. The secondary objective of this study is to evaluate prenatal and postnatal risk factors for acute kidney injury (AKI) in premature infants <30 weeks gestational age. The investigators will also compare various rates of complications including death, length-of-stay, and prolonged duration of mechanical ventilation, among others.

ELIGIBILITY:
Inclusion Criteria:

* Any neonate less than 30 weeks in gestational age
* Willingness and capacity of both adult parents/guardians to sign consent

Exclusion Criteria:

* An infant with known congenital anomalies of the kidney (i.e., grade 4 or 5 vesicoureteral reflux (VUR), posterior urethral valves, moderate or severe hydronephrosis, autosomal recessive polycystic kidney disease (ARPKD), bilateral renal agenesis or dysplasia)
* Age >30 weeks gestational age
* Age <24 weeks and <500 grams (will be excluded due to sensitivity of skin in this vulnerable population).
* Clinician's decision that NIRS is not suitable due to the patient's clinical condition

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Average NIRS Value (SrSO2) | Up to Day-of-life 7
  NIRS values measured as renal tissue oxygen saturation (SrSO2); measured continuously over first 7 days of life.

SECONDARY OUTCOMES:
Serum Creatinine Values | Day-of-life 1, Day-of-life 3, Day-of-life 7, Day-of-life 14
Average Urine Output | Up to Day of NICU Discharge (Approximately Day-of-life 7; subject to large individual variations)
Length-of-Stay in NICU | Day of NICU Discharge (Approximately Day-of-life 7; subject to large individual variations)
Duration of Non-Invasive Ventilation | Up to Day of NICU Discharge (Approximately Day-of-life 7; subject to large individual variations)
Duration of Mechanical Ventilation | Up to Day of NICU Discharge (Approximately Day-of-life 7; subject to large individual variations)

CONTACTS AND LOCATIONS:
Overall Officials: Sourabh Verma, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Jordan.nelson@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Jordan.nelson@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.